CLINICAL TRIAL: NCT02066857
Title: Use of Cast Versus Removable Splints for Minimally Displaced Distal Radius Fractures in Elderly Patients: A Prospective, Randomized Trial
Brief Title: Cast vs. Splints for Minimally Displaced Distal Radius Fractures in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Claudius Jarrett, Assistant Professor of Orthopaedics, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071060
Record Dates: First submitted 2014-02-14; First posted 2014-02-20 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Radius; Fracture, Lower or Distal End
Keywords: Wrist fracture; Radius fracture; Elderly; Splint; Cast
MeSH Terms: conditions — Fractures, Bone; Wrist Fractures; Radius Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic plaster or fiberglass cast group (Active Comparator): Patients will be randomized to receive a generic plaster or fiberglass cast for treatment of non-displaced distal radius fracture for 6 weeks.
  Interventions: Device: Cast made of generic plaster or fiberglass cast material
- Generic "off the shelf" removable splint group (Active Comparator): Subjects will be randomized and receive a generic "off the shelf" removable splint for treatment of non-displaced distal radius fracture for 6 weeks.
  Interventions: Device: Generic "off the shelf" removable splint

INTERVENTIONS:
Device: Cast made of generic plaster or fiberglass cast material — Patients will randomly receive a generic plaster or fiberglass cast for treatment of non-displaced distal radius fracture.
  Other Names: No brand name applicable.
  Arms: Generic plaster or fiberglass cast group
Device: Generic "off the shelf" removable splint — Patients will be randomized to receive a generic "off the shelf" removable splint for treatment of a non-displaced distal radius fracture.
  Other Names: No brand name applicable
  Arms: Generic "off the shelf" removable splint group

SUMMARY:
The purpose of this prospective randomized study is to add to the body of knowledge on the treatment of minimally displaced distal radius fractures in patients over 60 years of age. The investigators believe that treating minimally displaced distal radius fractures in people over 60 with a removable splint and early range of motion will provide greater patient satisfaction, fewer complications, and earlier functional returns to pre-injury for these patients compared to those treated with a short arm cast which immobilizes the limb for at least four weeks, and has been shown to lead to longer recovery and possible residual stiffness. The investigators hope to provide sufficient evidence in directing treatment that will give the most efficacious and the most satisfactory return of prior function to patients. Since distal radius fractures in the elderly are common because of poorer bone quality, the elderly proportion of the population is increasing, and controlling health costs is of current concern, answering the question of which treatment produces the best results for all these concerns is of increasing importance now.

ELIGIBILITY:
Inclusion Criteria:

1. Colles' Fracture - Distal radius fracture with dorsal angulation, apex volar (satisfies non-operative radiographic criteria before or after reduction
2. Isolated upper limb injury
3. No previous wrist fracture
4. Available for follow-up
5. Between 60 and 100 years of age

Exclusion Criteria:

1. Less than 60 years of age
2. Fractures that do not meet non-operative criteria or are deemed unstable by surgeon, subsequently requiring surgery after first clinic visit.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudius Jarrett, M.D., Principal Investigator — Emory University
Locations (1):
- Emory Orthopaedics and Spine Center, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Orthopaedic Fracture Clinic from April 2014 to November 2014.
Groups:
- Generic Plaster or Fiberglass Cast Group: Participants were randomized to receive a generic plaster or fiberglass cast for treatment of non-displaced distal radius fracture for 6 weeks.
- Generic "Off the Shelf" Removable Splint Group: Participants were randomized to receive a generic "off the shelf" removable splint for treatment of non-displaced distal radius fracture for 6 weeks.
Period: Overall Study
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group
Started | 1 | 4
Completed | 0 | 3
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Wrist Range of Motion (ROM)
Description: Wrist ROM will be assessed by a goniometer exam.
Time Frame: Baseline, Month 3
Population: Data for this outcome measure are not available for analysis.
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Mean Mayo Wrist Score
Description: The Mayo Wrist Score is a clinician-completed scoring system used to evaluate the level of functionality in the wrist, assessing pain, functional status (able to work), range of motion and grip strength. Total scores for functionality range from 0-100 and are categorized as follows: 90-100 indicates excellent, 80-90 indicates good, 60-80 indicates satisfactory, below 60 indicates poor. The assessment was completed at all study visits.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Of the 5 participants who were enrolled, data were analyzed for the 3 participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 3
units on a scale
  Baseline | 31.67 (16.07)
  Week 2 | 46.67 (20.21)
  Week 6 | 65 (10)
  Week 12 | 78.33 (2.89)

3. Primary Outcome: Change in Grip Strength
Description: Grip strength will be assessed by bilateral dynamometer testing.
Time Frame: Baseline, Month 3
Population: Data for this outcome measure are not available for analysis.
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Complication Rate
Description: The number of participants who experienced treatment related complications including the need for manipulation in the case of lost reduction.
Time Frame: Duration of Study (Up to 3 Months)
Population: Of the 5 participants who were enrolled, data were analyzed for the 3 participants who completed all study visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 3
Participants | 0

5. Primary Outcome: Mean Pain Score
Description: Pain will be assessed by a visual analog scale (VAS). Participants rate their pain level in a scale from 0 to 10; 0 representing "no pain" and 10 representing "the worst pain imaginable". The assessment was completed at all study visits.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Of the 5 participants who were enrolled, data were analyzed for the 3 participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 3
units on a scale
  Baseline | 6 (3.46)
  Week 2 | 3.66 (3.06)
  Week 6 | 1.67 (1.53)
  Week 12 | .33 (.58)

6. Secondary Outcome: Mean Disabilities of the Arm and Shoulder (DASH) Questionnaire Score
Description: The DASH questionnaire asks about symptoms as well as ability to perform certain activities. Scores range on a 0-100 scale. A higher score indicates greater disability.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Of the 5 participants who were enrolled, data were analyzed for the 3 participants who completed all study visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 3
units on a scale
  Baseline | 73.03 (23.53)
  Week 2 | 38.63 (27.11)
  Week 6 | 23.33 (22.50)
  Week 12 | 11.67 (16.07)

7. Secondary Outcome: Change in SF-12 QOL
Description: The SF-12 QOL is a self-administered measure asking views about participant's health and how well they are able to perform usual activities.
Time Frame: Baseline, Month 3
Population: No participants completed this survey as this outcome measure was removed from the protocol. No data were collected.
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collection for the duration of the study (2 years).
Arm/Group | Generic Plaster or Fiberglass Cast Group | Generic "Off the Shelf" Removable Splint Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
A small number of participants was analyzed due to limited enrollment and completion rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No